CLINICAL TRIAL: NCT05012176
Title: Episodic Future Thinking: An Interventional Pilot Study to Promote Weight Loss in Breast Cancer Survivors
Brief Title: An Episodic Future Thinking Intervention to Promote Weight Loss in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Sagar Sardesai, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-20408; NCI-2021-01597 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-07-13; First posted 2021-08-19 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Breast Ductal Carcinoma In Situ; Invasive Breast Carcinoma; Prognostic Stage 0 Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (EFT) (Experimental): Patients participate in EFT over 12 weeks, in which they will receive prompts via a guided smartphone application to engage in EFT in their daily lives. Patients are asked to recall future positive experiences to create text cues which vividly describes these experiences.
  Interventions: Behavioral: Behavioral Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (ERT) (Active Comparator): Patients participate in ERT over 12 weeks, in which they will receive prompts via a guided smartphone application to engage in ERT in their daily lives. Patients are asked to recall past positive experiences to create text cues which vividly describes these experiences.
  Interventions: Behavioral: Behavioral Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Participate in EFT
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm I (EFT)
Behavioral: Behavioral Intervention — Participate in ERT
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm II (ERT)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the use of an Episodic Future thinking Intervention to promote weight loss in breast cancer survivors. Obesity is associated with multiple negative health sequelae in breast cancer survivors. This includes an increased risk of cancer recurrence and mortality, multiple quality of life issues, and increased risk of co-morbidities.

Delay Discounting is a behavioral health economic target that refers to the "discounting" of a larger benefit in the future for a smaller, more immediate reward in the present. A high delay discounting rate is correlated with poor dietary choices and sedentary lifestyle. Episodic Future Thinking (EFT) simulates positive events that may occur in one's future, engaging the science of prospection. EFT decreases delay discounting rate, resulting in healthier diet choices and weight reduction. However, valuation of the future may impact cancer survivors differently due to adjusted mortality perception and cancer-related stress.

This study will determine the feasibility and preliminary efficacy of remotely delivered (smartphone application) EFT as a behavioral intervention for weight loss in breast cancer survivors. Implementation of EFT as a complementary approach to standard lifestyle interventions could lead to improvement in weight loss, food choice, and quality of life, thereby positively impacting overall health and longevity in cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the feasibility of the 12-week remotely delivered episodic future thinking (EFT) intervention.

SECONDARY OBJECTIVES:

I. To evaluate the impact of EFT compared to control (episodic recent thinking [ERT]) on weight loss and delay discounting (DD) in overweight and obese breast cancer survivors at 12 and 24 weeks.

II. To evaluate the baseline and 12 week change in:

IIa. Patient reported outcomes (PROs) measured by standard instruments: Patient Reported Outcomes Measurement Information System (PROMIS) scales 29 Profile version (v)2.1 (domains: physical function, social roles, fatigue, depression, anxiety, pain, sleep disturbance) and Global Health Short Form (general physical and mental health).

IIb. Insulin resistance (Homeostatic Model Assessment of Insulin Resistance [HOMA-IR]) and high-sensitivity C-reactive protein (hsCRP).

IIc. Diet quality, measured by Health Eating Index (HEI)-2015 on Vioscreen food frequency questionnaire (FFQ).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients participate in EFT over 12 weeks, in which they will receive prompts via a guided smartphone application to engage in EFT in their daily lives. Patients are asked to recall future positive experiences to create text cues which vividly describes these experiences.

ARM II: Patients participate in Episodic Recent Thinking (ERT; control arm) over 12 weeks, in which they will receive prompts via a guided smartphone application to engage in control thinking in their daily lives. Patients are asked to recall past positive experiences to create text cues which vividly describes these experiences.

After completion of study intervention, patients are followed up for an additional12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Breast cancer (BC) survivors (pathologically proven ductal carcinoma in situ or stage I-III invasive BC and completed primary breast surgery, radiation, chemotherapy >= 21 days prior to enrollment)
* Body mass index (BMI) >= 25 kg/m^2
* Endocrine and HER2- directed therapy is permitted
* Have access to a mobile electronic device
* Motivated to lose weight (readiness to change assessment)

Exclusion Criteria:

* Stage IV BC
* Have not completed definitive locoregional therapy (surgery +/- radiation therapy)
* Participating in another weight loss clinical trial
* Not able to speak and understand English
* Cognitive impairment which would interfere with performance of DD task or EFT procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Feasibility measured by Adherence | Up to 12 weeks
  A one-sample t-test will be used to evaluate adherence (average proportion of smartphone prompts participants open and attended to during the 12-week trial recorded by the web application)

SECONDARY OUTCOMES:
Change in total body weight | Up to 12 weeks
  Evaluated using a linear mixed effects model. The model will include baseline measure, timepoint (12 and 24 weeks), treatment assignment, and the timepoint by treatment interaction as fixed effects. A subject-level random effect will be included to account for the correlation of multiple measurements of the same individual.
Change in total body weight | Up to 24 weeks
  Evaluated using a linear mixed effects model. The model will include baseline measure, timepoint (12 and 24 weeks), treatment assignment, and the timepoint by treatment interaction as fixed effects. A subject-level random effect will be included to account for the correlation of multiple measurements of the same individual.
Change in delay discounting rate | Baseline to 12 weeks
  Evaluated using a linear mixed effects model. The model will include baseline measure, timepoint (12 weeks), treatment assignment, and the timepoint by treatment interaction as fixed effects. A subject-level random effect will be included to account for the correlation of multiple measurements of the same individual.
Change in delay discounting rate | Baseline to 24 weeks
  Evaluated using a linear mixed effects model. The model will include baseline measure, timepoint (24 weeks), treatment assignment, and the timepoint by treatment interaction as fixed effects. A subject-level random effect will be included to account for the correlation of multiple measurements of the same individual.

OTHER OUTCOMES:
Change in patient reported outcome (PRO) | Baseline to 12 weeks
  PRO measured by standard instruments: PROMIS® scales 29 Profile v2.1 (domains: physical function, social roles, fatigue, depression, anxiety, pain, sleep disturbance) and Global Health Short Form (general physical and mental health)
Change in Insulin Resistance | Baseline to 12 weeks
  Insulin Resistance will be measured by Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)
Change in quantity of serum high-sensitivity C-reactive protein | Baseline to 12 weeks
  Inflammatory Biomarker
Change in diet quality | Baseline to 12 weeks
  Measured by Health Eating Index 2015.

CONTACTS AND LOCATIONS:
Overall Officials: Sagar D Sardesai, MBBS MPH, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT05012176/ICF_000.pdf